CLINICAL TRIAL: NCT05802303
Title: Safety and Efficacy of Transdermal Estrogen (Gel) Versus Oral Estrogen for Endometrial Preparation in Down-regulated Frozen Embryo Transfer (FET) Cycles-An Open-label Multi Centric Randomized Controlled Trial
Brief Title: Estrogen (Gel)Transdermal vs Oral Estrogen for Endometrial Preparation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As per institutional protocol unable to recruit adequate number of patients
Sponsor: Indira IVF Hospital Pvt Ltd (Other)
Responsible Party: Principal Investigator, Dr Vipin Chandra, Chief Clinical Lab Operations, Indira IVF Hospital Pvt Ltd
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIHPL-UDR/RCT/002_2022
Record Dates: First submitted 2023-02-21; First posted 2023-04-06 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Frozen Embryo Transfer; Infertility, Female
Keywords: Transdermal Estrogen; FET; Oral Estrogen; IVF/ICSI
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant
Masking Description: All cases undergoing frozen embryo transfer with own or donor gametes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transdermal Gel (Active Comparator): In the Estradiol gel group patients will be administered transdermal Estradiol gel (17-beta Estradiol gel 0.06%)
  Interventions: Drug: 17-beta Estradiol gel 0.06% w/w(ESTOGEL.Intas pharma)
- Oral Estradiol (Other): In the Oral Estradiol group, all women will be given oral Estradiol valerate tablets
  Interventions: Drug: Estradiol Hemihydrate(Estrabet Tablet, abbott pharma)

INTERVENTIONS:
Drug: 17-beta Estradiol gel 0.06% w/w(ESTOGEL.Intas pharma) — In the Estradiol gel group patients will be administered transdermal Estradiol gel (17-beta Estradiol gel 0.06% w/w) 2 puffs thrice a day (each application contains 1.25 mg with 0.75 mg of the drug).
  Arms: Transdermal Gel
Drug: Estradiol Hemihydrate(Estrabet Tablet, abbott pharma) — In the oral Estradiol group, all women will be given 2 mg of Estradiol valerate tablets, one tablets thrice a day within 30 days of injection triptorelin depot. Endometrial assessment will be performed on D10 of HRT. Please see the flow diagram (in the annexure) for details.
  Arms: Oral Estradiol

SUMMARY:
The goal of this randomized study trial is to comparing transdermal estradiol gel and oral estradiol for endometrial preparation in the Frozen Embryo Transfer Cycle. The main question[s] it aims to answer is: • Can Transdermal estrogen (gel) can be equally efficacious as compared to oral estrogen in hormone replacement FET (HRT- FET) cycles ? The Transdermal gel would have the added benefit of a higher patient comfort with fewer side effects and a better safety profile. Participants planned for Frozen embryo transfer will undergo H-P-O axis suppression on previous cycle D21 of menses with gonadotropin-releasing hormone(GnRH) agonist depot preparation (Inj. Decapeptyl 3.75 mg) IM . The study will compare Transdermal E2 gel with Oral E2 tabs. The patients will be randomized into an oral and gel group, and all patients will participate only once in the study.

DETAILED DESCRIPTION:
Estrogen priming is essential for the induction of progesterone receptors and to build endometrial thickness, both of which play an important role in regulating endometrial receptivity . Different routes of Estrogen administration are oral (tablets), transdermal (patch/gel), and vaginal (tablets).

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients aged 23-35 years.
* BMI 18.5 to 29.9 kg/m2.
* A normal uterine cavity assessed by 3D ultrasound (USG)/hysteroscopy.
* Patients who underwent IVF/ICSI and who have cryopreserved their embryos.
* Those receiving donor oocytes or donor embryos.
* Patients undergoing hormonal replacement frozen embryo transfer (HRT-FET) cycles with GnRH agonist suppression.
* Embryo Transfers of good quality embryos -2/3/4/5 AA, AB, BA(As per Gardner Grading System).

Exclusion Criteria:

* Preimplantation Genetic Testing for Aneuploidies (PGT-A) cycles.
* Patients who had a FET performed in natural or stimulated cycles.
* Patients who had more than 2 failed transfers due to thin endometrium.
* Patients having uterine anomalies.
* Known cases of adenomyosis and endometriosis.
* Underlying cardiac/renal/hepatic/thromboembolic disorders, h/o anxiety or depression.
* E2 >50 pg./ml, P4 > 1 ng/ml and on D2 of menses.
* On D2 scan presence of a cyst or a dominant follicle.
* Patients with a history of recurrent 1st-trimester abortions.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All women planned for Frozen embryo transfer
Enrollment: 172 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness (ET) | 14 to 21 days after start of estrogen
  Average endometrial thickness achieved on day 14 of HRT

SECONDARY OUTCOMES:
Cycle cancelation rate | 21 days after starting HRT
  Number of cycles cancelled before embryo transfer × 100
Average E2 consumption | On 1 day of embryo transfer
  Total E2 consumed till embryo transfer
Implantation rates (IR) | 4 weeks + 2 weeks after embryo transfer
  The number of gestational sacs observed by transvaginal ultrasound at the 6th gestational week per the number of embryos transferred.
Clinical pregnancy rates (CPR) | 4 weeks + 2 weeks after embryo transfer
  Detection of a foetal heartbeat on transvaginal ultrasound at the 6th gestational week per embryo transfer cycle
Miscarriage rates (MR) | Within 20 weeks of gestation
  Number of spontaneous pregnancy losses in which a gestational sac was previously observed (before gestation week <20 weeks) per 100 clinical pregnancy .
Patient satisfaction score | on 1 day of embryo transfer
  It is measured using visual analogue scale(VAS) score

OTHER OUTCOMES:
Undesirable side effects between both the groups | Till 12 weeks of pregnancy
  Symptoms like rash, itching ,burning, thromboembolic event

CONTACTS AND LOCATIONS:
Locations (1):
- Indira IVF Hospital Private Limited, Udaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers after publication of primary results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After 6 months of publication of primary results

REFERENCES:
- [Background] Bourdon M, Santulli P, Kefelian F, Vienet-Legue L, Maignien C, Pocate-Cheriet K, de Mouzon J, Marcellin L, Chapron C. Prolonged estrogen (E2) treatment prior to frozen-blastocyst transfer decreases the live birth rate. Hum Reprod. 2018 May 1;33(5):905-913. doi: 10.1093/humrep/dey041. PMID 29529202
- [Background] Scheffer JB, Scheffer BB, Aguiar APS, Franca JB, Lozano DM, Fanchin R. A comparison of the effects of three different estrogen used for endometrium preparation on the outcome of day 5 frozen embryo transfer cycle. JBRA Assist Reprod. 2021 Feb 2;25(1):104-108. doi: 10.5935/1518-0557.20200059. PMID 32991118
- [Background] Corroenne R, El Hachem H, Verhaeghe C, Legendre G, Dreux C, Jeanneteau P, Descamps P, May-Panloup P, Bouet PE. Endometrial preparation for frozen-thawed embryo transfer in an artificial cycle: transdermal versus vaginal estrogen. Sci Rep. 2020 Jan 22;10(1):985. doi: 10.1038/s41598-020-57730-3. PMID 31969591
- [Background] Devroey P, Pados G. Preparation of endometrium for egg donation. Hum Reprod Update. 1998 Nov-Dec;4(6):856-61. doi: 10.1093/humupd/4.6.856. PMID 10098476
- [Background] Garimella S, Karunakaran S, Gedela DR. A prospective study of oral estrogen versus transdermal estrogen (gel) for hormone replacement frozen embryo transfer cycles. Gynecol Endocrinol. 2021 Jun;37(6):515-518. doi: 10.1080/09513590.2020.1793941. Epub 2020 Jul 15. PMID 32666854
- [Background] Ranisavljevic N, Raad J, Anahory T, Grynberg M, Sonigo C. Embryo transfer strategy and therapeutic options in infertile patients with thin endometrium: a systematic review. J Assist Reprod Genet. 2019 Nov;36(11):2217-2231. doi: 10.1007/s10815-019-01576-w. Epub 2019 Sep 9. PMID 31502111
- [Background] Paulson RJ. Hormonal induction of endometrial receptivity. Fertil Steril. 2011 Sep;96(3):530-5. doi: 10.1016/j.fertnstert.2011.07.1097. PMID 21880274
- [Background] Shahrokh Tehraninejad E, Kabodmehri R, Hosein Rashidi B, Jafarabadi M, Keikha F, Masomi M, Hagholahi F. Trans dermal estrogen (oestrogel) for endometrial preparation in freeze embryo transfer cycle: An RCT. Int J Reprod Biomed. 2018 Jan;16(1):51-56. PMID 29675488